CLINICAL TRIAL: NCT02521649
Title: An Open, Dose-ranging, Multicenter Study to Determine the Antibody Response to G17DT and Its Safety and Tolerability in the Treatment of Patients With Gastric Cancer
Brief Title: Dose-ranging Study to Evaluate Antibody Response to G17DT in Patients With Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Collaborators: Clinical Project Services (Unknown); MPS Research Unit (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC2
Record Dates: First submitted 2015-05-15; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; G17DT; PAS; Insegia; Gastrimmune
MeSH Terms: conditions — Stomach Neoplasms | interventions — gastrin immunogen

ARMS (5):
- 10µg, Stage I-III (Experimental): 10µg/0.2 mL dose of G17DT administered at Weeks 0,2, and 6 with an option of a 125µg/0.1 mL dose of G17DT administered at Week 12 based on measured antibody titer.
  Interventions: Drug: G17DT
- 100µg, Stage I-III (Experimental): 100µg/0.2 mL dose of G17DT administered at Weeks 0,2, and 6 with an option of a 125µg/0.1 mL dose of G17DT administered at Week 12 based on measured antibody titer.
  Interventions: Drug: G17DT
- 250µg, Stage I-III (Experimental): 250µg/0.2 mL dose of G17DT administered at Weeks 0,2, and 6 with an option of a 125µg/0.1 mL dose of G17DT administered at Week 12 based on measured antibody titer.
  Interventions: Drug: G17DT
- 100µg, Stage IV (Experimental): 100µg/0.2 mL dose of G17DT administered at Weeks 0,2, and 6 with an option of a 125µg/0.1 mL dose of G17DT administered at Week 12 based on measured antibody titer.
  Interventions: Drug: G17DT
- 250µg, Stage IV (Experimental): 250µg/0.2 mL dose of G17DT administered at Weeks 0,2, and 6 with an option of a 125µg/0.1 mL dose of G17DT administered at Week 12 based on measured antibody titer.
  Interventions: Drug: G17DT

INTERVENTIONS:
Drug: G17DT
  Other Names: Gastrimmune, Insegia, PAS

SUMMARY:
An open, dose-ranging, multiple dose, multi-centre study in patients with Stage I-III or Stage IV gastric cancer. Twelve patients in each of 5 treatment groups were to receive three injections at weeks 0, 2 and 6 with provision for a single booster injection in an extension study period.

ELIGIBILITY:
Inclusion Criteria:

Stage I-III Criteria-

* Patients aged 18 years or over who had had a macroscopically curative resection for gastric adenocarcinoma.
* Absence of metastatic disease evident from:

  * physical examination
  * the most recent chest X-ray
  * abdominal CT or ultrasound scan
* Life expectancy of at least 3 months
* WHO performance status of 0 to 1
* Written informed consent given

Stage IV Criteria-

* Patients aged 18 years or over with Stage IV gastric cancer: carcinoma with the primary tumour invading the adjacent structures and/or involvement of more than 15 regional lymph nodes and/or distant metastases
* Life expectancy of at least 3 months
* WHO performance status of 0 to 2
* Written informed consent given

Exclusion Criteria:

* History of other malignant disease except non-melanomatous skin cancer or in situ carcinoma of the uterine cervix Recurrent gastric cancer following previous surgery Presence of metastatic disease: peritoneal deposits or involved lymph nodes outside the limit of resection
* Previous use, concomitant use or anticipated use in the period of the study, of any anti-cancer therapies
* Concomitant use of immunosuppressants, including systemic (ie oral or injected) corticosteroids
* Females who were pregnant, planning to become pregnant or lactating
* Patients who were taking part in another study involving an investigational or licensed drug or device in the three months preceding enrolment or during this study
* Previous G17DT treatment
* Haematological indicators:

  * Haemoglobin <10.0g/dl
  * White blood cell count <4.0 x 109/l
  * Platelets <100 x 109/l

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 1998-09; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
Measurable Antibody Titer | Up to Week 12

SECONDARY OUTCOMES:
Overall Survival from date of randomization to death or end of study | Up to Last Patient Last Visit, January 2001
  Patients were scheduled to attend follow-up visits every four weeks after completion of the 12-week core period of the study and to continue until the patient was discharged from the study or declined further follow-up.
Injection Site Reaction | Through Week 12
  A physical examination for the presence of an abcess at the injection site was performed on each patient to assess tolerability to treatment at every posttreatment visit from Week 0 to Week 12.